CLINICAL TRIAL: NCT03139604
Title: GRAVITAS-301: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of Itacitinib or Placebo in Combination With Corticosteroids for the Treatment of First-Line Acute Graft-Versus-Host Disease
Brief Title: GRAVITAS-301: A Study of Itacitinib or Placebo in Combination With Corticosteroids for Treatment of Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 39110-301; 2017-000538-78 (EudraCT Number)
Record Dates: First submitted 2017-05-02; First posted 2017-05-04 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Acute graft-versus-host disease; Janus kinase (JAK) inhibitor; itacitinib; corticosteroids; allogeneic hematopoietic stem cell transplant (allo-HSCT)
MeSH Terms: conditions — Graft vs Host Disease | interventions — itacitinib; INCB039110; Prednisone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Itacitinib (Experimental): Itacitinib plus corticosteroids
  Interventions: Drug: Itacitinib; Drug: Prednisone; Drug: Methylprednisolone
- Placebo (Placebo Comparator): Matching placebo plus corticosteroids
  Interventions: Drug: Placebo; Drug: Prednisone; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Itacitinib — Itacitinib at the protocol-defined dose administered orally once daily (QD) plus corticosteroids.
  Other Names: INCB039110
  Arms: Itacitinib
Drug: Placebo — Matching placebo tablets administered orally once daily (QD) plus corticosteroids.
  Arms: Placebo
Drug: Prednisone — Oral prednisone may be used to begin standard corticosteroid background treatment at the investigator's discretion, at a dose equivalent to methylprednisolone 2 mg/kg per day.
  Other Names: Deltasone; Prednicot; predniSONE Intensol; Rayos; Sterapred; Sterapred DS
Drug: Methylprednisolone — Methylprednisolone 2 mg/kg IV daily (or prednisone equivalent) or at a dose appropriate for the severity of disease as background treatment.
  Other Names: Medrol; Medrol Dosepak; Solu-Medrol

SUMMARY:
The purpose of this study is to evaluate itacitinib or placebo in combination with corticosteroids as first-line treatment of participants with Grade II to IV acute graft-versus-host disease (aGVHD).

ELIGIBILITY:
Inclusion Criteria:

* Has undergone 1 allo-HSCT from any donor (related or unrelated with any degree of HLA matching) and any donor source (bone marrow, peripheral blood stem cells, or cord blood) for a hematologic malignancy or disorder. Recipients of myeloablative and reduced-intensity conditioning regimens are eligible.
* Clinically suspected Grade II to IV aGVHD as per MAGIC criteria, occurring after allo-HSCT and any GVHD prophylaxis regimen.
* Evidence of myeloid engraftment. Use of growth factor supplementation is allowed.
* Serum creatinine ≤ 2.0 mg/dL or creatinine clearance ≥ 40 mL/min measured or calculated by Cockroft Gault equation.
* Willing to avoid pregnancy or fathering children.
* Able to give written informed consent and comply with all study visits and procedures.
* Able to swallow and retain oral medication.

Exclusion Criteria:

* Has received more than 1 allo-HSCT.
* Has received more than 2 days of systemic corticosteroids for aGVHD.
* Presence of GVHD overlap syndrome.
* Presence of an active uncontrolled infection.
* Known human immunodeficiency virus infection.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation.
* Participants with evidence of relapsed primary disease, or participants who have been treated for relapse after the allo-HSCT was performed.
* Any corticosteroid therapy for indications other than GVHD at doses > 1 mg/kg per day methylprednisolone (or prednisone equivalent) within 7 days of randomization.
* Severe organ dysfunction unrelated to underlying GVHD, including:

  * Cholestatic disorders or unresolved veno-occlusive disease of the liver.
  * Clinically significant or uncontrolled cardiac disease.
  * Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
* Currently breast feeding.
* Received JAK inhibitor therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
* Treatment with any other investigational agent, device, or procedure within 21 days (or 5 half-lives, whichever is greater) of enrollment.
* Any medical complications or conditions that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Morariu-Zamfir, MD, Study Director — Incyte Corporation
Locations (129):
- United States (49):
  - University of California, San Diego (UCSD) - Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - University of Florida (UF) - Division of Hematology & Oncology, Gainesville, Florida
  - University of Miami - Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Lutheran General Hospital - Oncology Specialists SC, Park Ridge, Illinois
  - Indiana University (IU) Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplant, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Tulane University Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - John Theurer Cancer Center At Hackensack UMC, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Northwell Health, Lake Success, New York
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest Baptist Medical Center - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Oncology Hematology in Cincinnati, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University (OSU), Columbus, Ohio
  - University of Oklahoma - Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Methodist Healthcare Foundation, Memphis, Tennessee
  - Sarah Cannon Research Institute, LLC (SCRI), Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Transplant Institute, San Antonio, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
- St Vincents Hospital Sydney Limited, Darlinghurst, Australia
- Ordensklinikum Linz GmbH Elisabethinen, Linz, Austria
- Belgium (8):
  - ZNA Stuivenberg, Antwerp
  - General Hospital Sint-Jan Brugge-Oostend, Bruges
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent (UZG), Ghent
  - Jessa Ziekenhuis, Hasselt
  - Hopital universitaire du Sart Tilman de Liege, Liège
  - AZ Delta, Roeselare
- UHKT Prague - Institute of Hematology and Blood Transfusion, Prague, Czechia
- Helsinki University Central Hospital, Helsinki, Finland
- France (8):
  - CHU Amiens Picardie - Hopital Sud, Amiens
  - CHRU de Lille-Hopital Claude Huriez, Lille
  - Hotel Dieu Hospital - Hematologie, Nantes
  - Hopital Saint Louis, Paris
  - Hopital Haut Leveque - CHU Bordeaux - Maladies du sang, Pessac
  - Hopital de Hautepierre, Strasbourg
  - Institut Claudius Regaud-Universitaire du Cancer Toulouse Oncopol, Toulouse
  - CHU de Nancy, Vandœuvre-lès-Nancy
- Germany (7):
  - Universitaet zu Koln - Universitaetsklinikum Koeln (Uniklinik Koeln), Cologne
  - University Clinic Carl Gustav Carus, Technical University Dresden, Dresden
  - Universitatsklinikum Freiburg - Klinik fur Innere Medizin I, Freiburg im Breisgau
  - Universitatsklinikum Hamburg - Eppendorf, Hamburg
  - Universitaetsklinikum Leipzig, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg, Mainz
  - UKGM Marburg Innere Medizin: Haematologie Onkolog, Marburg
- General Hospital of Thessaloniki G. Papanikolaou - Hematology Department, Chortiatis, Greece
- Israel (4):
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center Ein Karem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (17):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII, Bergamo
  - C.T.M.O. Ospedale Roberto Binaghi ATS Cagliari, Cagliari
  - Azienda Ospedaliero Universitaria (AOU) Policlinico - Vittorio Emanuele - Presidio Ospedaliero Ferrarotto Alessi, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Clinica Ematologica CTA, Ospedale "San Gerardo" di Monza, Monza
  - Casa di Cura La Maddalena, Palermo
  - Fondazione IRCCS Policlinco San Matteo, Pavia
  - Presidio Ospedaliero Pescara, Pescara
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli Ospedali Riuniti, Reggio Calabria
  - Azienda Unità Sanitaria Locale di Reggio Emilia, Reggio Emilia
  - University of Rome La Sapienza, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. Città della Salute e della Scienza di Torino, Torino
  - SOC Clinica Ematologica, Azienda Ospediero-Universitaria di Udine, Udine
- Auckland District Health Board, Auckland, New Zealand
- Poland (2):
  - Centrum Onkologii- Instytut w Gliwicach, Gliwice
  - Klinika Transplantacji Komorek Krwiotworczych - Instytut Hematologii i Transfuzjologii, Warsaw
- Portugal (3):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil EPE (IPO-Lisboa), Lisbon
  - Centro Hospitalar Lisboa Norte - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Seoul National University Hospital, Seoul, South Korea
- Spain (16):
  - Hospital de la Santa Creu i Sant Pau - Servei de Hematologia Clinica, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, Barcelona
  - Complejo Hospitalario Universitario de Granada - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (3):
  - Universtity Hospital Basel - Haematology, Basel
  - Hopitaux Universitaires de Geneve, Geneva
  - Universitaetsspital Zuerich - Klinik fuer Haematology, Zurich
- China Medical University Hospital, Taichung, Taiwan
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Hammersmith Hospital, London
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pratta M, Paczesny S, Socie G, Barkey N, Liu H, Owens S, Arbushites MC, Schroeder MA, Howell MD. A biomarker signature to predict complete response to itacitinib and corticosteroids in acute graft-versus-host disease. Br J Haematol. 2022 Aug;198(4):729-739. doi: 10.1111/bjh.18300. Epub 2022 Jun 11. PMID 35689489
- [Derived] Zeiser R, Socie G, Schroeder MA, Abhyankar S, Vaz CP, Kwon M, Clausen J, Volodin L, Giebel S, Chacon MJ, Meyers G, Ghosh M, Deeren D, Sanz J, Morariu-Zamfir R, Arbushites M, Lakshminarayanan M, Barbour AM, Chen YB. Efficacy and safety of itacitinib versus placebo in combination with corticosteroids for initial treatment of acute graft-versus-host disease (GRAVITAS-301): a randomised, multicentre, double-blind, phase 3 trial. Lancet Haematol. 2022 Jan;9(1):e14-e25. doi: 10.1016/S2352-3026(21)00367-7. PMID 34971577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 128 investigative sites in 19 different countries.
Pre-assignment Details: A total of 498 participants were screened for this study, of which 59 participants were screen failures and 439 participants were randomized to treatment.
Groups:
- Itacitinib Plus Corticosteroids: Itacitinib was administered at a starting dose of 200 mg orally once daily QD (2 × 100 mg tablets) in combination with steroids i.e. methylprednisolone 2 mg/kg IV daily (or prednisone equivalent) or at a dose that is appropriate for the severity of the disease.
- Placebo Plus Corticosteroids: Matching placebo was administered orally once daily QD in combination with steroids i.e. methylprednisolone 2 mg/kg IV daily (or prednisone equivalent) or at a dose that is appropriate for the severity of the disease.
Period: Overall Study
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Started | 219 | 220
Completed | 0 (Participants were considered to have completed the study if they dies or discontinued study treatment for any reason) | 0 (Participants were considered to have completed the study if they dies or discontinued study treatment for any reason)
Not Completed | 219 | 220
Not completed — Other | 7 | 3
Not completed — Withdrawal by Subject | 16 | 17
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 65 | 67
Not completed — Study Terminated by Sponsor | 122 | 127
Not completed — Final EOS data missing due to COVID-19 restrictions that affected on-site monitoring | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids | Total
Number analyzed (Participants) | 219 | 220 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.53) | 54.0 (12.96) | 53.8 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 91 | 173
  Male | 137 | 129 | 266
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 17 | 22 | 39
  Not Hispanic or Latino | 167 | 169 | 336
  Not Reported | 17 | 14 | 31
  Unknown | 12 | 9 | 21
  Other | 6 | 5 | 11
  Missing | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  White/Caucasian | 196 | 194 | 390
  Black/African-American | 8 | 5 | 13
  Asian | 4 | 4 | 8
  American-Indian/Alaska Native | 0 | 2 | 2
  Other | 10 | 11 | 21
  Missing | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Based on Center for International Blood and Marrow Transplant Research (CIBMTR) Response Index
Description: Defined as the percentage of participants demonstrating a complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: Day 28
Population: Full Analysis Set (FAS) Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
Percentage of Participants | 74.0 [67.6 to 79.7] | 66.4 [59.7 to 72.6]
Statistical Analysis 1: Comparison: Itacitinib Plus Corticosteroids vs Placebo Plus Corticosteroids; binomial distribution; Test type: Other; p = 0.0782, Cochran-Mantel-Haenszel — Not adjusted for multiplicity with interim and final analyses; Odds Ratio (OR) = 1.45, 95% CI 2-sided [0.959 to 2.204]

2. Secondary Outcome: Nonrelapse Mortality
Description: Defined as the percentage of participants who died due to causes other than malignancy relapse.
Time Frame: Month 6,9,12 and 24
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants
  6 Months | 36 | 37
  9 Months | 46 | 45
  12 Months | 51 | 52
  24 Months | 56 | 52

3. Secondary Outcome: Duration of Response
Description: Defined as the interval from first response until GVHD progression or death.
Time Frame: Baseline through 30-35 days after end of treatment, total particpation expected to average 24 months
Population: Full Analysis Set (FAS) Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
days | 587 [513 to NA] — Upper bound is not estimable | NA [NA to NA] — Not Estimable

4. Secondary Outcome: Cmax of Itacitinib When Administered in Combination With Corticosteroids
Description: Defined as maximum observed plasma concentration.
Time Frame: Protocol-defined timepoints up to Day 28
Population: All subjects who receive at least 1 dose of study drug and provide at least 1 plasma sample after study drug administration will be considered as potential PK evaluable subjects. The data presented is from Day 7.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Itacitinib Plus Corticosteroids
Number analyzed (Participants) | 162
nM | 796 (642)

5. Secondary Outcome: Cmin of Itacitinib When Administered in Combination With Corticosteroids
Description: Defined as minimum observed plasma concentration.
Time Frame: Protocol-defined timepoints up to Day 28
Population: All subjects who receive at least 1 dose of study drug and provide at least 1 plasma sample after study drug administration will be considered as potential PK evaluable subjects. The data presented is from Day 7 as this is more representative of true steady state. Day 28 is positively biased as non responders are withdrawn from study by D28.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Itacitinib Plus Corticosteroids
Number analyzed (Participants) | 62
nM | 72.5 (121)

6. Secondary Outcome: Tmax of Itacitinib When Administered in Combination With Corticosteroids
Description: Defined as time to maximum plasma concentration.
Time Frame: Protocol-defined timepoints up to Day 28
Population: as for outcome 4
Measure: Median (Full Range); unit: hrs
Arm/Group | Itacitinib Plus Corticosteroids
Number analyzed (Participants) | 62
hrs | 2.1 [0.83 to 5.3]

7. Secondary Outcome: AUC of Itacitinib When Administered in Combination With Corticosteroids
Description: Defined as area under the concentration-time curve.
Time Frame: Protocol-defined timepoints up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nM*h
Arm/Group | Itacitinib Plus Corticosteroids
Number analyzed (Participants) | 62
nM*h | 6720 (6210)

8. Secondary Outcome: CL/F of Itacitinib When Administered in Combination With Corticosteroids
Description: Defined as oral dose clearance.
Time Frame: Protocol-defined timepoints up to Day 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Itacitinib Plus Corticosteroids
Number analyzed (Participants) | 62
L/h | 104 (76.7)

9. Secondary Outcome: Time to Response
Description: Defined as the interval from treatment initiation to first response
Time Frame: End of Study, total particpation expected to average 24 months
Population: Full Analysis Set (FAS) Population who were responders
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 195 | 185
days | 9.9 (6.25) | 10.1 (5.37)

10. Secondary Outcome: Relapse Rate of Malignant and Nonmalignant Hematologic Disease
Description: Defined as the proportion of subjects whose underlying hematologic disease relapses
Time Frame: Randomization through end of Study, study duration expected to average 24 months
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: percentage
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 217 | 220
percentage | 12.4 | 11.4

11. Secondary Outcome: Malignancy Relapse-related Mortality Rate
Description: Defined as the proportion of subjects whose malignancy relapses and has a fatal outcome.
Time Frame: Randomization through end of Study, study duration expected to average 24 months
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: percentage
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
percentage | 6.4 | 7.7

12. Secondary Outcome: Failure-free Survival
Description: Defined as the proportion of subjects who are still alive, have not relapsed, have not required additional therapy for aGVHD, and have not demonstrated signs or symptoms of chronic graft-versus-host disease (cGVHD)
Time Frame: 6 months from randomization
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: proportion of participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
proportion of participants | 44.29 | 40.00

13. Secondary Outcome: Overall Survival (OS)
Description: Defined as the interval from study enrollment to death due to any cause.
Time Frame: End of Study up to approximately 24 months
Population: Full Analysis Set (FAS) Population
Measure: Median (Full Range); unit: days
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
days | 365 [1 to 867] | 348.5 [1 to 827]

14. Secondary Outcome: Number of Treatment-emergent Adverse Events With INCB39110
Description: Adverse events reported for the first time or worsening of a pre-existing event after the first dose of study treatment
Time Frame: 30-35 days after end of treatment, approximately 24 months
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 215 | 216
participants | 208 | 214

15. Secondary Outcome: Incidence Rate of Secondary Graft Failure
Description: Defined as > 95% recipient cells any time after engraftment with no signs of relapse, OR retransplantation because of secondary neutropenia (< 0.5 × 109/L) and/or thrombocytopenia (< 20 × 109/L) within 2 months of transplantion
Time Frame: Randomization through end of Study, study duration expected to average 24 months
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants | 2 | 0

16. Secondary Outcome: Proportion of Subjects Who Discontinue Corticosteroids
Description: Average and cumulative corticosteroid dose usage will be calculated and proportion of subjects discontinuing corticosteroids will be tabulated
Time Frame: Days 28, 56, 100, and 180
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 215 | 216
participants
  Day 28 | 3 | 3
  Day 56 | 16 | 11
  Day 100 | 39 | 45
  Day 180 | 39 | 45

17. Secondary Outcome: Proportion of Subjects Who Discontinue Immunosuppressive Medications
Description: Summary statistics of subjects discontinuing immunosuppressive medications will be calculated
Time Frame: Days 56 and 100
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants
  Day 56 | 12 | 10
  Day 100 | 11 | 8

18. Secondary Outcome: Incidence Rate of aGVHD Flares
Time Frame: up to day 100
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants | 42 | 48

19. Secondary Outcome: Incidence Rate of cGVHD
Time Frame: Days 180 and 365
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants
  Day 180 | 25 | 36
  Day 365 | 43 | 58

20. Secondary Outcome: Objective Response Rate
Time Frame: Days 14, 56 and 100
Population: Full Analysis Set (FAS) Population
Measure: Number; unit: participants
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids
Number analyzed (Participants) | 219 | 220
participants
  Day 14 | 170 | 160
  Day 56 | 138 | 124
  Day 100 | 92 | 96

ADVERSE EVENTS:
Time Frame: 30 days after last dose approximately up to 24 months
Groups:
- Total: Total
Arm/Group | Itacitinib Plus Corticosteroids | Placebo Plus Corticosteroids | Total
All-Cause Mortality (participants affected / at risk) | 69/215 | 69/216 | 138/431
Serious Adverse Events (participants affected / at risk) | 133/215 | 131/216 | 264/431
Other Adverse Events (participants affected / at risk) | 207/215 | 206/216 | 413/431
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib Plus Corticosteroids (N=215) | Placebo Plus Corticosteroids (N=216) | Total (N=431)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5) | 7 (7)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 3 (3) | 4 (4)
Acute graft versus host disease in skin (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 5 (5) | 13 (13)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 3 (3) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 5 (5)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Bacteraemia (Infections and infestations) | 0 (0) | 4 (4) | 4 (4)
Bacterial sepsis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3)
Bronchopulmonary aspergillosis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 4 (4) | 0 (0) | 4 (4)
Cytomegalovirus infection (Infections and infestations) | 2 (2) | 3 (3) | 5 (5)
Cytomegalovirus infection reactivation (Infections and infestations) | 6 (6) | 1 (2) | 7 (8)
Cytomegalovirus viraemia (Infections and infestations) | 5 (5) | 5 (5) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 10 (11) | 13 (15) | 23 (26)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Enterovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Escherichia infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Escherichia sepsis (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
Fatigue (General disorders) | 2 (2) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 8 (10) | 15 (18)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 3 (3) | 4 (4)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 3 (3) | 6 (6) | 9 (9)
Graft versus host disease in lung (Immune system disorders) | 0 (0) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 9 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 4 (4)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Limbic encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Microangiopathy (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
Mucormycosis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 5 (5)
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 6 (6)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 11 (12) | 13 (15) | 24 (27)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pneumonia influenzal (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 1 (1) | 2 (2) | 3 (3)
Pseudomonal sepsis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 4 (4)
Pyrexia (General disorders) | 15 (19) | 10 (10) | 25 (29)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 1 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) | 8 (8)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory tract infection fungal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 6 (6) | 11 (11)
Septic shock (Infections and infestations) | 2 (2) | 6 (6) | 8 (8)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 4 (4) | 5 (5)
Steroid diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 1 (1) | 5 (5)
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 9 (9)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 6 (6)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Toxoplasmosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1) | 4 (5)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral haemorrhagic cystitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4) | 7 (7)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Adenoviral hepatitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Bartter's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Bullous oedema of the bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Clostridium test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Disseminated aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 1 (1) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 3 (3) | 3 (3)
Enterococcus test positive (Investigations) | 1 (1) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Fungal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Klebsiella test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rotavirus test positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Sinusitis aspergillus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Sinusitis fungal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal subdural haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Venoocclusive liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib Plus Corticosteroids (N=215) | Placebo Plus Corticosteroids (N=216) | Total (N=431)
Abdominal pain (Gastrointestinal disorders) | 26 (32) | 26 (28) | 52 (60)
Acute kidney injury (Renal and urinary disorders) | 11 (13) | 21 (23) | 32 (36)
Alanine aminotransferase increased (Investigations) | 30 (39) | 21 (23) | 51 (62)
Anaemia (Blood and lymphatic system disorders) | 63 (80) | 54 (66) | 117 (146)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (24) | 18 (19) | 41 (43)
Aspartate aminotransferase increased (Investigations) | 23 (37) | 13 (18) | 36 (55)
Asthenia (General disorders) | 12 (15) | 19 (19) | 31 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (20) | 21 (25) | 38 (45)
Blood alkaline phosphatase increased (Investigations) | 12 (14) | 16 (19) | 28 (33)
Blood cholesterol increased (Investigations) | 16 (19) | 11 (13) | 27 (32)
Blood creatinine increased (Investigations) | 25 (27) | 19 (20) | 44 (47)
Constipation (Gastrointestinal disorders) | 25 (27) | 21 (22) | 46 (49)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (35) | 42 (54) | 74 (89)
Cytomegalovirus infection (Infections and infestations) | 16 (20) | 10 (12) | 26 (32)
Cytomegalovirus infection reactivation (Infections and infestations) | 26 (35) | 24 (26) | 50 (61)
Cytomegalovirus viraemia (Infections and infestations) | 34 (38) | 26 (30) | 60 (68)
Decreased appetite (Metabolism and nutrition disorders) | 24 (26) | 23 (26) | 47 (52)
Diarrhoea (Gastrointestinal disorders) | 42 (48) | 43 (60) | 85 (108)
Dizziness (Nervous system disorders) | 23 (24) | 17 (19) | 40 (43)
Dry eye (Eye disorders) | 18 (18) | 17 (19) | 35 (37)
Dry mouth (Gastrointestinal disorders) | 14 (15) | 18 (24) | 32 (39)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 (31) | 15 (19) | 43 (50)
Dysuria (Renal and urinary disorders) | 17 (18) | 8 (8) | 25 (26)
Fall (Injury, poisoning and procedural complications) | 20 (22) | 21 (23) | 41 (45)
Fatigue (General disorders) | 28 (32) | 37 (54) | 65 (86)
Gamma-glutamyltransferase increased (Investigations) | 11 (11) | 7 (8) | 18 (19)
Headache (Nervous system disorders) | 20 (21) | 32 (39) | 52 (60)
Hyperglycaemia (Metabolism and nutrition disorders) | 47 (56) | 50 (57) | 97 (113)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (11) | 16 (23) | 25 (34)
Hypertension (Vascular disorders) | 46 (52) | 31 (35) | 77 (87)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 31 (33) | 27 (34) | 58 (67)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (13) | 23 (26) | 35 (39)
Hypocalcaemia (Metabolism and nutrition disorders) | 16 (17) | 20 (21) | 36 (38)
Hypokalaemia (Metabolism and nutrition disorders) | 40 (51) | 35 (43) | 75 (94)
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 (46) | 21 (28) | 48 (74)
Hyponatraemia (Metabolism and nutrition disorders) | 16 (27) | 22 (27) | 38 (54)
Hypophosphataemia (Metabolism and nutrition disorders) | 14 (18) | 11 (13) | 25 (31)
Insomnia (Psychiatric disorders) | 22 (23) | 25 (26) | 47 (49)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 23 (24) | 19 (20) | 42 (44)
Nausea (Gastrointestinal disorders) | 38 (47) | 33 (45) | 71 (92)
Neutropenia (Blood and lymphatic system disorders) | 36 (57) | 40 (59) | 76 (116)
Oedema (General disorders) | 7 (7) | 16 (16) | 23 (23)
Oedema peripheral (General disorders) | 53 (55) | 53 (61) | 106 (116)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (15) | 13 (13) | 27 (28)
Platelet count decreased (Investigations) | 38 (45) | 22 (25) | 60 (70)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (14) | 17 (24) | 30 (38)
Pyrexia (General disorders) | 34 (44) | 31 (38) | 65 (82)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 14 (15) | 20 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 73 (87) | 69 (77) | 142 (164)
Tremor (Nervous system disorders) | 27 (28) | 19 (21) | 46 (49)
Upper respiratory tract infection (Infections and infestations) | 17 (25) | 17 (19) | 34 (44)
Urinary tract infection (Infections and infestations) | 15 (15) | 17 (19) | 32 (34)
Vomiting (Gastrointestinal disorders) | 23 (26) | 25 (27) | 48 (53)
Anxiety (Psychiatric disorders) | 17 (17) | 13 (13) | 30 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 12 (16) | 18 (22)
Dysgeusia (Nervous system disorders) | 11 (12) | 2 (3) | 13 (15)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 13 (13) | 23 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11) | 20 (20)
Epstein-Barr virus infection reactivation (Infections and infestations) | 11 (11) | 6 (6) | 17 (17)
Hypotension (Vascular disorders) | 16 (16) | 11 (11) | 27 (27)
Leukopenia (Blood and lymphatic system disorders) | 6 (8) | 11 (14) | 17 (22)
Nasopharyngitis (Infections and infestations) | 7 (8) | 11 (12) | 18 (20)
Neuropathy peripheral (Nervous system disorders) | 6 (6) | 11 (11) | 17 (17)
Neutrophil count decreased (Investigations) | 15 (18) | 9 (11) | 24 (29)
Oral candidiasis (Infections and infestations) | 11 (13) | 11 (11) | 22 (24)
Pancytopenia (Blood and lymphatic system disorders) | 11 (11) | 6 (6) | 17 (17)
Pneumonia (Infections and infestations) | 5 (6) | 11 (11) | 16 (17)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 3 (3) | 14 (14)
Vision blurred (Eye disorders) | 7 (7) | 12 (13) | 19 (20)
Weight decreased (Investigations) | 11 (11) | 8 (10) | 19 (21)
White blood cell count decreased (Investigations) | 12 (18) | 10 (11) | 22 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement

DOCUMENTS (2):
  • Study Protocol (2018-08-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03139604/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT03139604/SAP_001.pdf